CLINICAL TRIAL: NCT00470522
Title: A Canadian Multicenter, Randomized, Double-Blind Placebo-Controlled Study of Methotrexate and Folic Acid in Systemic Lupus Erythematosus: A Phase III Trial.
Brief Title: Study of Methotrexate in Lupus Erythematosus
Acronym: SMILE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAS Grant 95072
Record Dates: First submitted 2007-05-02; First posted 2007-05-07 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: methotrexate; folic acid; systemic lupus erythematosus; steroid
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Methotrexate; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methotrexate and folic acid

SUMMARY:
The treatment of systemic lupus erythematosus (SLE) has been aimed at decreasing mortality and morbidity because the etiology of the disease is unknown. The general aim of this multicentre randomized placebo-controlled trial of low dose intermittent methotrexate with folic acid is to establish whether methotrexate shows efficacy and safety in controlling disease activity in SLE and preventing flares in disease activity or development of end-organ damage. A second aim will be to document the steroid sparing effect of methotrexate in SLE. A Third aim will be to measure toxicity and utility of methotrexate with folic acid and to perform effectiveness and utility analyses.

DETAILED DESCRIPTION:
SLE is a chronic systemic autoimmune and inflammatory disease. Approximately 65% of patients develop SLE between 16 and 55 years of age, and it is 8-10 times more common in women. Overall prevalence is estimated at 40-50 per 100,000 individuals in the US. SLE typically includes periods of remission and flares. Systemic manifestation of SLE includes fatigue, fever, arthralgia, weight loss, and skin rash. Disease progression is variable and unpredictable from one individual to the next. Treatment is aimed at preventing damage due to inflammation of the involved tissues. Death occur primarily from severe systemic infections and renal insufficiency. Futhermore, patients with long-standing SLE on chronic steroid use may succumb from atherosclerotic complications such as myocardial infarction.

The mainstay of treatment of acute disease manifestations is steroids, in particular,prednisone. Once started, it is difficult to reduce or stop treatment without new flares or severe steroid withdrawal. Longitudinal studies in SLE cannot dissociate morbidity caused by the disease from that caused by prolonged steroid use.

Specific Objectives:

1. To measure the efficacy, safety and tolerance of methotrexate with folic acid compared to placebo with folic acid.
2. To measure the steroid-sparing effects of methotrexate in SLE
3. To perform a cost-effectiveness and a cost-utility analysis of methotrexate with folic acid using generic and disease specific health status measures.

Qualification for the study:

Once written informed consent is obtained, subjects will have a screening visit and laboratory evaluations performed to determine if they qualify for the study. A patient is enrolled in the study once all eligibility criteria are met. No change in dosage of prednisone, NSAIDs or plaquenil will be allowed between screening and qualifying visits.

Assignment of the treatment:

After qualifying for the study, subjects will be randomly assigned to receive one of two treatments: placebo with folic acid 2.5 mg/day except on the day they take methotrexate or placebo, or methotrexate at doses described below with folic acid 2.5 mg/day except on the day whem methotrexate or placebo is taken.

Treatment period: All patients will receive study medication (placebo or methotrexate) for at least 12 months. If the patient is on steroid, every effort will be done to taper prednisone according to a schedule. One flare requiring increase dose of steroid higher than baseline (dose determined by local investigator) will be allowed. If a second flare occurs, it will mean stopping the trial. There will be an open phase at the end of the trial during which those responding favorably to methotrexate and those on placebo will be offered to either continue or start methotrexate for 6 months.

Drug formulation, route of administration, dosage and duration:

Methotrexate:

Patients will be randomly assigned to receive either methotrexate or MTX-placebo (except formulation of the placebo consists of 44.00 mg of lactose, 31.00 mg of maize starch, 2.5 mg of pregelatinized starch, 0.20 mg of polysorbate 80, 1.00 mg of riboflavin, 20.70 mg of microcrystalline cellulose, 1.50 mg of magnesium stearate and small quantities of purified water and sodium hydroxide 1N). It will be given orally. Each tablet contains 2.5 mg of methotrexate or equivalent color, size and shape-matched placebo. Subject will be given 3 MTX tablets, 2.5 mg increment or an equivalent number of MTX-placebo. Subjects ill be given 3 MTX tablets, of 2.5 mg.increment or an equivalent number of MTX-placebo tablets to take all together once a week for 12 months. If the patient does not have symptoms, signs or laboratory evidence of toxicity after 2 weeks, MTX will be increased by 2.5 mg per 8 week intervals until maximal does of 0.25 mg/kg/week or 20 mg/week is achieved. In the absence of toxicity, MTX will be continued at that does or the maximal tolerated dose for 12 months.Dose will be adjusted according to the guidelines for MTX does reduction for toxicity. At the end of the blinded period, those patients who have completed the 12 months blinded study, who have benefited from MTX with FA and want to continue or try it (for those who were on placebo) will be offered to continue into an open-label trial of MTX with FA.

Folic Acid:

Folic acid at a dose of 2.5 mg/day for 6 days/week will be given early to all patients. Folic acid will not be given on the day the methotrexate or placebo is taken. folic acid is a vitamin which has no known anti-inflammatory or immunosuppressive activity at this dose and no known toxicity.

Guidelines for methotrexate dose reduction for toxicity:

Strict guidelines have been defined for the adjustment of the dose of MTX or placebo. In each participating centre, the physician who will review the laboratory tests and adjust the dose will be different from the physician who will assess disease activity and clinical response to the treatment. Both physicians will be blinded to the study drug, but this is done as supplementary precaution to protect blinding should blood tests suggest that a patient is on placebo or on MTX.

Open-label trial:

Patient who terminate from the study prematurely will not be eligible to receive further treatment with MTX in this follow-up study. The open trial model will be modeled on the protocol except for the blinding. Patients who were receiving MTX will be offered continuation of the drug with the same surveillance mechanism for an extra 6 months. Those who were receiving MTX-placebo will be offered to try MTX. At the end of this 6 months, the open label trial will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* men and women with diagnosis of SLE
* 18 years and above
* negative pregnancy test for female subjects of child-bearing age and must accept not to attempt to get pregnant during the period of the study
* Subject with active disease as defined by SLAM of at least 8
* SLICC/ACR damage index of less or equal to 15
* Subject must be on stable does of NSAIDs, prednisone, or antimalarial (chloroquine sulfate or hydroxychloroquine) at least 4 weeks preceding the study
* subjects can be under other medications as long as condition or treatment will not interfere with the experimental medications and assessments
* must understand either French or English and can give written informed consent

Exclusion Criteria:

* previous history of hypersensitivity or intolerance to methotrexate or folic acid
* total SLAM of less than 8 or total SLICC/ACR score of more than 15.
* history of medical non-compliance or inability to comply with instructions
* subject who have received intra-articular or intramuscular corticosteroids in the four weeks prior to study entry.
* clinically significant acute or chronic liver disease with the exception of autoimmune liver disease
* alcohol use in excess of 2 ounces of 100 proof liquor or its equivalent/week
* insulin requiring diabetes mellitus with morbid obesity
* renal impairment such that the serum creatinine is more than or equal to 175 umol/I (SI units) or 2.0 mg/dl
* interstitial lung disease as defined by an abnormal chest x-ray or decrease diffusion capacity (DLCO < 70% of predicted) without evidence of pulmonary hypertension.
* WBC count ,3,000/ cubic mm. and/or platelet count ,80,000/ cubic mm.
* prior use of methotrexate to treat SLE
* use of sulfa drugs that may potentiate the folate antagonistic effects of MTX
* non-steroidal anti-inflammatory drugs will be allowed throughout the trial unless there is evidence of renal failure or other contra-indications to these drugs. Their con-comitant use with MTX is routine in patients with rheumatoid arthritis.
* use of another cytotoxic or immunosuppressive drug such as cyclophosphamide, azathioprine, chlorambucil, cyclosporin or trimetoprime currently or in the preceding 6 months.
* current participation in any other drug trial or participation in such a trial in the previous one month.
* serologic evidence of infection with HIV
* biologic potential for pregnancy and not utilizing effective means of contraception
* recently (less than 6 months) diagnosed malignancy
* vitamin B12 deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 1995-06; Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
SLAM - Systemic Lupus Activity Measure | at one year
Daily dose of prednisone | at one year

SECONDARY OUTCOMES:
SLICC DI - Systemic Lupus International Collaborating Clinic Damage Index | at one year
SF-36 - Short Form 36 | at one year
SLEDAI - Systemic Lupus Erythematosus Disease Activity Index | at one year

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. Fortin, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada